CLINICAL TRIAL: NCT00750217
Title: Transfer From Methadone to Buprenorphine Maintenance Treatment Using Buprenorphine Patches: A Study on Practicability With Patients Maintained With Daily Dosages Between 60mg and 100mg Methadone.
Brief Title: Transfer From Methadone to Buprenorphine Maintenance Treatment Using Buprenorphine Patches
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Psychiatric University Hospital, Zurich (Other)
Responsible Party: Stohler Rudolf MD, Psychiatric University Hospital, Zurich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-54/2007
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2008-09-10 (Estimated); Status verified 2008-08

CONDITIONS: Heroin Addiction
Keywords: transfer methadone buprenorphine patch heroin addiction
MeSH Terms: conditions — Heroin Dependence | interventions — Administration, Sublingual; Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Buprenorphine patch and sublingual tablets — Buprenorphine patch: 35 micro grams per hour 12 to 48 hours after last methadone intake.
  Buprenorphine sublingual tablets: 2mg 48 and 60 hours after last methadone intake; 8mg 72 and 84 hours after last methadone intake; 8mg 96, 102 and 109 hours after last methadone intake.
  Other Names: Transtec (buprenorphine patch); Subutex (buprenorphine sublingual tablets)

SUMMARY:
Buprenorphine is an important alternative to methadone in the maintenance treatment of heroin addiction. Transfer from methadone to buprenorphine requires a reduction of daily methadone dosage below 30 mg to avoid withdrawal after the first buprenorphine intake. The study hypothesis states that the transfer from a daily methadone dosage between 60 mg and 100 mg to buprenorphine can be carried out without withdrawal using buprenorphine patches (35 micro grams per hour) within 12 to 48 hours after last methadone intake.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years
* Methadone maintenance treatment for at least 3 months preceding the study
* Daily methadone dosage between 60mg amd 100mg
* Sufficient knowledge of German language
* Ability to give informed consent

Exclusion Criteria:

* Daily methadone dosage below 60mg amd over 100mg
* Prescribed use of benzodiazepines over 30 mg equivalent to diazepam
* Misuse or dependence of alcohol and/or GHB/GBL
* Pregnant or breast-feeding women
* Known intolerance of buprenorphine
* Somatic diseases interfering with the study plan

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-02 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Short Opiate Withdrawal Scale | 14 days

SECONDARY OUTCOMES:
Heroin use | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Stohler, MD, Study Director — Psychiatric University Hospital; Lukas Boesch, PhD, Study Chair — Psychiatirc University Hospital
Locations (1):
- Psychiatric University Hospital, Zurich, Canton of Zurich, Switzerland